CLINICAL TRIAL: NCT00938262
Title: An Open-label, Three-treatment, Three-period, One-sequence, Crossover Study to Evaluate the Effect of Ketoconazole and Rifampicin on the Pharmacokinetics of Fimasartan in Healthy Male Volunteers
Brief Title: A Study to Evaluate the Effect of Ketoconazole and Rifampicin on the Pharmacokinetics of Fimasartan in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Choi, Director, Boryung Pharmaceutical Co., Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A657-BR-CT-105
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan; Ketoconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fimasartan, Ketoconazole, Rifampicin (Experimental)
  Interventions: Drug: Fimasartan, Ketoconazole, Rifampicin

INTERVENTIONS:
Drug: Fimasartan, Ketoconazole, Rifampicin — Fimasartan (1 day)
  Ketoconazole (3 days) Ketoconazole + Fimasartan (1 day)
  Rifampicin (9 days) Rifampicin + Fimasartan (1 day)

SUMMARY:
To evaluate the effect of ketoconazole and rifampicin on the pharmacokinetics of fimasartan.

ELIGIBILITY:
Inclusion Criteria:

* age: 20 - 45 years
* sex: male
* body weight: greater than 55 kg
* written informed consent

Exclusion Criteria:

* known allergy to Fimasartan, ketoconazole and rifampicin
* existing cardiac or hematological diseases
* existing hepatic and renal diseases
* existing gastrointestinal diseases
* acute or chronic diseases which could affect drug absorption or metabolism
* history of any serious psychological disorder
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day 3 month ago
* participation in a clinical trial during the last 2 months prior to the start of the study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Cmax, AUClast, AUCinf, CL/F, Tmax, t1/2 | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 32, (48, 56) h